CLINICAL TRIAL: NCT06834477
Title: The Influence of Structural and Microenvironmental Abnormalities in the Olfactory Cleft on Olfactory Function in Patients With Chronic Rhinosinusitis
Brief Title: Impact of Structural and Microenvironmental Abnormalities in Olfactory Cleft on Olfaction in CRS
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dawei Wu, Associate Researcher, Peking University Third Hospital
Other Study IDs: 9059102
Record Dates: First submitted 2025-02-06; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Rhinosinusitis (CRS)
Keywords: olfactory cleft; olfactory dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Mucus from the olfactory cleft and biopsy specimens from the posterior end of the superior turbinate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CRS admitted for endoscopic sinus surgery
  Interventions: Other: Computed Tomography
- healthy controls undergoing surgery for the deviated septum
  Interventions: Other: Computed Tomography

INTERVENTIONS:
Other: Computed Tomography — low-dose CT is taken
  Other Names: collection of superior turbinate biopsy specimens; collection of olfactory cleft mucus

SUMMARY:
The purpose of this research is to investigate the impact of structural abnormalities and microenvironmental changes in the olfactory cleft on olfactory function in patients with chronic rhinosinusitis (CRS). It sought to elucidate the complex relationships among structural abnormalities, microenvironmental changes, and inflammatory factors contributing to olfactory dysfunction through a multidimensional assessment encompassing imaging, aerodynamics, biomarker , and histopathology analysis.

DETAILED DESCRIPTION:
Olfactory dysfunction (OD) is a critical symptom among patients with CRS, affecting up to 83% of individuals with the condition. Currently, it is considered that the inflammation in olfactory cleft is a central factor contributing to both conductive and sensorineural OD in patients with CRS. Inflammation in the olfactory cleft could impair olfaction by altering the mucosal and mucus microenvironment thereby causing damage to the olfactory neuroepithelium, by physically impeding delivery of odorant-containing air to the olfactory cleft, or a combination of both mechanisms.

Existing studies mainly focus on isolated mechanisms, such as inflammation-induced physical obstruction or injury of olfactory epithelium. However, limited research has explored how structural abnormalities and microenvironmental changes in the olfactory cleft might interact to contribute to olfactory dysfunction. This research aimed to evaluate the relationship between structural abnormalities and microenvironmental changes in the olfactory cleft and their impact on olfactory function in patients with CRS using a multidimensional approach integrating imaging, pathology, and functional analysis.

This is a retrospective study. Patients with CRS admitted for endoscopic sinus surgery (n = 70) and healthy controls undergoing surgery for the deviated septum (n = 10) were included. All the participants had undergone:

1. Clinical assessment of olfactory function and quality of life

   1. Olfactory measurements had been conducted preoperatively using the Sniffin' Sticks Test to evaluate olfactory threshold (OT), olfactory discrimination (OD), olfactory identification (OI), and the overall composite scores (TDI). A TDI score > 30.75, 16-30.75, and ≤ 15 indicates normosmia, hyposmia, and anosmia, respectively.
   2. The 22-item Sino-Nasal Outcome Test (SNOT-22) had been administered to evaluate patient-reported subjective outcomes.
   3. The Questionnaire of Olfactory Disorders Negative Statements (QOD-NS) was utilized to assess the olfactory-specific quality of life.
   4. The visual analog scale（VAS）for olfaction was employed to measure patients' self-reported olfaction.
2. Evaluation of structural abnormalities and patency of the olfactory cleft

   Computed tomography scans were obtained in every participant. The anterior boundary of OC is defined by the anterior attachment of the middle turbinate; the posterior boundary corresponding to the anterior face of the sphenoid sinus; the lateral boundaries are defined as the attachment of the middle and/or superior turbinate laterally and the nasal septum medially. The olfactory cleft is further divided into anterior and posterior, divided by the anterior end of the superior turbinate. The olfactory cleft opacification is defined as the normal airway filled with a value representing soft tissue and /or presence of close contact between the nasal turbinates and the nasal septum. The opacification percentage in the anterior olfactory cleft is calculated using the lower margin of the middle turbinate and the cribriform plate as the vertical boundaries. The opacification percentage in the posterior olfactory cleft is calculated using the lower margin of the superior turbinate and the cribriform plate as the vertical boundaries. The olfactory cleft opacifications were graded on a scale of 0-4 by the ratio of the opacified area to the whole area of the corresponding region of the olfactory cleft, with 0 (no opacification), 1 (25%), 2 (25%-50%), 3 (50%-75%), and 4 (>75%). Then we evaluated:
   1. The original version of olfactory cleft CT score, calculated as the sum of the anterior and posterior olfactory cleft opacification scores, ranged from 1 to 8.
   2. The modified version of olfactory cleft CT score: CT scores for unilateral olfactory cleft, including the anterior and posterior regions, specifically the left anterior, left posterior, right anterior, and right posterior olfactory cleft, as well as their total sum. Additionally, a more detailed assessment is performed by recording whether opacification is present at the apex and the middle-lower portion of each olfactory cleft subregion. Each subregion is further divided into anterior, middle, and posterior areas, with each area being independently assessed. A score of 1 is assigned if opacification is observed, and 0 if absent.

   To further quantify the impact of olfactory cleft obstruction on olfactory airflow, this study employs three-dimensional modeling and computational fluid dynamics (CFD) analysis of the nasal cavity based on CT imaging data of sinuses. The air flow, velocity, pressure, and air flow ratio in the olfactory cleft were obtained by the hydrodynamics analysis method.
3. Evaluation of the mucus and mucosal microenvironment in the olfactory cleft

   1. Patients with CRS were categorized into two clinical phenotypes, CRS with nasal polyps (CRSwNP) and CRS without nasal polyps (CRSsNP), based on histology and physical examination.
   2. To investigate the inflammatory phenotypes of CRS, hematoxylin and eosin (H&E) staining were performed to identify the predominant inflammatory cell types within the lamina propria. Patients with CRS were divided into eosinophilic CRS and non-eosinophilic CRS. The eosinophilic phenotype of CRS was defined when the frequency of tissue eosinophils exceeded 10% of the total infiltrating cells per high-power field.
   3. Olfactory cleft mucus was collected to quantify the level of olfactory cleft mucus galectin-10 and eosinophil-derived neurotoxin (EDN) using commercial human enzyme-linked immunosorbent assay kits. Th1/Th2-related cytokines, including IL-2, IL-4, IL-5, IL-6, IFN-γ, TNF, and IL-10, were detected using a flow cytometry-based bead array (CBA) capture assay.
   4. Olfactory cleft mucosal specimens were collected from the anterior portion of the superior turbinate using a through-cut forceps during surgery for immunohistochemical analysis of olfactory marker protein (OMP), to evaluate the expression levels of mature olfactory neurons.

ELIGIBILITY:
Inclusion Criteria for patient group:

1. Diagnosed with CRS based on the diagnostic criteria of the EPOS guideline.
2. Provision of signed and dated informed consent form.
3. Patients with CRS admitted to the hospital awaiting endoscopic sinus surgery.

Inclusion Criteria for control group:

1. Healthy controls undergoing surgery for the deviated septum.
2. Provision of signed and dated informed consent form.

Exclusion Criteria for patient group:

1. Those who have taken oral glucocorticoids, antibiotics, anti-leukotrienes, and antihistamines within four weeks.
2. Patients who have had prior sinus surgery.
3. Patients with fungal sinusitis, inverted papilloma, or other nasal diseases.
4. Patients with a diagnosis of immune suppression or suspicion of malignancy that may be affecting the nose/paranasal sinuses.
5. Patients who are mentally or physically unable to perform olfactory tests

Exclusion Criteria for control group:

1. Patients with nasal polyps, sinusitis, nasal cavity tumors and other diseases.
2. Patients with hyposmia or anosmia.
3. Patients with diagnosed neurodegenerative disease.
4. Patients who are mentally or physically unable to perform olfactory tests.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical patients were recruited from the Department of Otolaryngology at Peking University Third Hospital in clinic.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-14 (Estimated); Primary Completion 2027-03-14 (Estimated); Study Completion 2027-03-14 (Estimated)

PRIMARY OUTCOMES:
Sniffin Sticks Test | Immediately before surgery
  The test consists of odorous rods that are presented to the patient's nose. It consists of 3 parts different, with 3 sets of corresponding sticks: an olfactory threshold test, an olfactory discrimination test and an olfactory identification test.
  The final TDI score, out of 48, is the sum of the olfactory threshold, discrimination and identification scores.

SECONDARY OUTCOMES:
The 22-item Sino-Nasal Outcome Test (SNOT-22) | Immediately before surgery
Visual analog scale（VAS）for olfaction | Immediately before surgery
  numerical rating scale from 0 (no smell) to 10 (perfect smell)
The Questionnaire of Olfactory Disorders Negative Statements (QOD-NS) | Immediately before surgery
  The QOD-NS comprises 17 negatively phrased statements, each rated on a scale from 0 (disagree) to 3 (agree), yielding a maximum score of 51. Higher QOD-NS scores indicate a poorer quality of life.
The original version of olfactory cleft CT score | during routine preoperative CT imaging
The modified version of olfactory cleft CT score | during routine preoperative CT imaging
Airflow velocity in the olfactory cleft | Immediately after CT scans
  one of the airflow parameters in the olfactory cleft that can be obtained by CFD analysis
Mass flowrate in the olfactory cleft | Immediately after CT scans
  One of the airflow parameters in the olfactory cleft that can be obtained by CFD analysis
Airflow ratio in the olfactory cleft | Immediately after CT scans
  one of the airflow parameters in the olfactory cleft that can be obtained by CFD analysis. The airflow ratio was calculated as the mass flowrate through the OC relative to the total airflow rate through the nasal cavity.
The level of eosinophil-derived neurotoxin, galectin-10 and otherTh1/Th2-related cytokines in olfactory cleft mucus | Immediately after surgery
  The levels of galectin-10 and eosinophil-derived neurotoxin (EDN) in olfactory cleft mucus were measured by commercial human enzyme-linked immunosorbent assay kits. Th1/Th2-related cytokines, including IL-2, IL-4, IL-5, IL-6, IFN-γ, TNF, and IL-10, were detected using a flow cytometry-based bead array (CBA) capture assay.
Clinical phenotypes classification：CRS with nasal polyps (CRSwNP) or CRS without nasal polyps (CRSsNP) | During preoperative physical and imaging examinations
Histopathological phenotypes classification: eosinophilic CRS or non-eosinophilic CRS | Immediately after surgery
  Hematoxylin and eosin (H&E) staining are performed to identify the predominant inflammatory cell types within the lamina propria. Patients with CRS were divided into eosinophilic CRS and non-eosinophilic CRS.
Immunohistochemical staining of olfactory marker protein (OMP) in olfactory epithelium | Immediately after surgery
  The OMP is a kind of biomarker for mature olfactory sensory neurons. This parameter may indicate the inflammation-induced neurological damage in olfactory epithelium.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otolaryngology Head and Neck Surgery, Peking University Third Hospital, Beijing, People's Republic of China, Beijing, Haidian District, China

IPD SHARING:
Plan to Share IPD: No
We will decide whether to share the individual participant data after the study.